CLINICAL TRIAL: NCT04393051
Title: BARICIVID-19 STUDY: MultiCentre, Randomised, Phase IIa Clinical Trial Evaluating Efficacy and Tolerability of Baricitinib as add-on Treatment of In-patients With COVID-19 Compared to Standard Therapy
Brief Title: Baricitinib Compared to Standard Therapy in Patients With COVID-19
Acronym: BARICIVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Francesco Menichetti, Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BARICIVID-19
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; SARS-CoV 2; SARS Pneumonia
Keywords: baricitinib; invasive ventilation; safety; pneumonia; SARS-CoV2; Covid-19
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Phase II randomized clinical trial to evaluate the efficacy and safety of baricitinib in patients with SARS-CoV2 pneumonia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAR group (Experimental): Patients who will be assigned (after a computerized randomization) to the BAR group will. receive baricitinib as adjunctive therapy.
  Baricitinib will be administered at 4 mg daily via oral route for 14 days as add-on therapy or 2 mg daily via oral route (eGFR between 30 and 60 ml/min and for patients with age >75 years old) for 14 days as add-on therapy
  Interventions: Drug: Baricitinib Oral Tablet
- Control group (No Intervention): Patients in the control group will continue to receive standard therapy.

INTERVENTIONS:
Drug: Baricitinib Oral Tablet — Baricitinib will be administered by oral route at different dosages according to age and kidney function. The drug will be administered for 14 days, unless occurrence of discontinuation criteria.
  Arms: BAR group

SUMMARY:
There is urgent need of an effective therapy for Covid-19. To date, the best treatment of SARS-CoV-2 infection is unknown. Baricitinib has been identified as potential treatment for 2019-nCoV acute respiratory disease, because of its immunomodulating and hypothesized antiviral activity.

This is a multicenter randomized clinical trial that aims to evaluate the efficacy and safety of baricitinib in patients with SARS-CoV2 pneumonia. Patients will be randomized to receive or not baricitinib as adjunctive therapy. All patients will continue to receive the ongoing standard therapy: chloroquine/idrossichloroquine and low-molecular weight heparin (LMWH) eventually associated with ritonavir/lopinavir or darunavir/ritonavir will be allowed for all included patients.

The primary endpoint measure is the efficacy of baricitinib in reducing the number of patients requiring invasive ventilation after 7 and 14 days of treatment.

Secondary endpoints will be mortality rates and toxicity of baricitinib.

DETAILED DESCRIPTION:
There is urgent need of an effective therapy for Covid-19. To date, the best treatment of SARS-CoV-2 infection is unknown. Multiple strategies have been proposed and several randomized clinical trials are ongoing. Recently, data extracted from scientific literature by machine learning suggested a potential role of baricitinib, a Janus kinases (JAKs) inhibitor, that induces an anti-inflammatory effect and a dose dependent inhibition of IL-6. This drug is currently approved for the treatment of rheumatoid arthritis. However, it has been suggested that this drug may act against SARS-CoV-2 by inhibiting of the AP2-associated protein kinase 1 (AAK1), a regulator of the endocytosis pathway exploited by SARS-CoV-2 to infect lung cells through binding with ACE2. Disruption of AAK1 might interrupt the passage of the virus into cells and also the intracellular assembly of virus particles.

The aim of this study is to evaluate the efficacy and safety of baricitinib in patients with SARS-CoV2 pneumonia.

This is a multicenter randomized controlled clinical trial for evaluating efficacy, safety and tolerability of baricitinib added to the usual care treatments in comparison with the usual care treatments, enrolling patients with COVID-19 /SARS-CoV2 pneumonia.

The primary endpoint measure is the efficacy of baricitinib in reducing the number of patients requiring invasive ventilation after 7 and 14 days of treatment.

Secondary endpoints will be: mortality rate after 14- and 28-days from randomization; time to invasive mechanical ventilation (days); time to independence from non-invasive mechanical ventilation (days); time to independence from oxygen therapy (days); time to improvement in oxygenation for at least 48 hours (days); length of hospital stay (days); length of ICU stay (days); instrumental response (pulmonary echography); toxicity of baricitinib.

All patients included in the study will be treated with the usual care treatments. One group will receive baricitinib by oral route, while the control group will continue the usual care treatments. In the intervention group, baricitinib will be administered at the dosage of 4 mg daily by oral route for 14 consecutive days. For patients with eGFR between 30 and 60 ml/min and for patients with age >75 years old, the dosage will be half a tablet a day (2 mg/day) for 14 days.

Inclusion criteria are the following

* Any gender
* Age > 18 years on day of signing informed consent
* Informed written consent for participation in the study
* Virological diagnosis of SARS-CoV-2 infection (real-time PCR)
* Hospitalized due to clinical instrumental diagnosis of pneumonia
* Oxygen saturation at rest in ambient air ≤93% or P/F ratio <250
* Able to be administered by oral route drugs
* Patients who receive O2 therapy or who need non-invasive mechanical ventilation
* In case of female patients at childbearing potential, they should agree to use highly effective methods of birth control at least till 7 days after the termination of the treatments

Exclusion criteria are the following:

* Known hypersensitivity to Baricitinib or its excipients
* Patients with Creatinine Clearance < 30 ml/min
* Patients with active Tuberculosis (TBC)
* Patients with known HBV or HCV infection
* Patients with deep vein thrombosis (DVP) or Pulmonary Embolism (PE)
* Patients with ALT or AST> 5 times the upper limit of the normality
* Neutrophils <1000/mmc
* Platelets <50.000/mmc
* Hb< 8g/dl
* Bowel diverticulitis or perforation
* Patients who receive invasive mechanical ventilation
* Documented bacterial infection at time of randomization
* Patients with "do not resuscitate order"
* Patients receiving immunosuppressants or anti-rejection drugs
* Pregnancy or breastfeeding

All patients, required by the assignment arm, will continue to receive therapy already in place, including that for Sars-CoV2 infection. Chloroquine/idrossichloroquine and low-molecular weight heparin (LMWH) eventually associated with ritonavir/lopinavir or darunavir/ritonavir will be allowed for all included patients.

For the duration of the study, the following will not be allowed:

* the concomitant use of IL-1 or IL-6 blockers, JAK inhibitors and TNF inhibitors
* the start of the steroid in the two weeks of study. The steroid will be continued if the patient already takes steroid at the time of admission

Intervention:

Intervention arm:

* BARICITINIB 4 mg daily via oral route for 14 days as add-on therapy
* BARICITINIB 2 mg daily via oral route (eGFR between 30 and 60 ml/min and for patients with age >75 years old) for 14 days as add-on therapy

Control arm:

- patients in the control group will continue to receive standard therapy

Sample size calculation:

Expected 7-days and 14-days invasive ventilation (P0):30% Auspicated 7-days and 14-days invasive ventilation (P1):12% Statistical power: 80% Bilateral alpha error: 5% Sample size needed: 63 patients for each group (126 total patients)

The statistical analysis plan will be developed and finalized before database lock and will describe the participant populations to be included in the analyses, and procedures for accounting for missing, unused, and spurious data.

An intention-to-treat (ITT) and per-protocol (PP) analysis will be performed on randomized patients and on the overall population, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age > 18 years on day of signing informed consent
* Informed written consent for participation in the study
* Virological diagnosis of SARS-CoV-2 infection (real-time PCR)
* Hospitalized due to clinical instrumental diagnosis of pneumonia.
* Oxygen saturation at rest in ambient air ≤93% or P/F ratio <250
* Able to be administered by oral route drugs
* Patients who receive O2 therapy or who need non-invasive mechanical ventilation
* In case of female patients at childbearing potential, they should agree to use highly effective methods of birth control at least till 7 days after the termination of the treatments

Exclusion Criteria:

* Known hypersensitivity to Baricitinib or its excipients
* Patients with Creatinine Clearance < 30 ml/min
* Patients with active Tuberculosis (TBC)
* Patients with known HBV or HCV infection
* Patients with deep vein thrombosis (DVP) or Pulmonary Embolism (PE)
* Patients with ALT or AST> 5 times the upper limit of the normality
* Neutrophils <1000/mmc
* Platelets <50.000/mmc
* Hb< 8g/dl
* Bowel diverticulitis or perforation
* Patients who receive invasive mechanical ventilation
* Documented bacterial infection at time of randomization
* Patients with "do not resuscitate order"
* Patients receiving immunosuppressants or anti-rejection drugs
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Need of invasive mechanical ventilation | after 7 and 14 days of treatment
  Reduction of the number of patients requiring invasive ventilation

SECONDARY OUTCOMES:
Mortality | 14- and 28-days from randomization
  Proportion of any cause deaths
Time to invasive mechanical ventilation | 30 days
  Days from randomization to invasive mechanical ventilation
Time to independence from non-invasive mechanical ventilation | 30 days
  Days from randomization to independence from non-invasive mechanical ventilation
Time to independence from oxygen therapy | 30 days
  Days from randomization to independence from oxygen therapy
Time to improvement in oxygenation for at least 48 hours | 30 days
  Days from randomization to improvement in oxygenation for at least 48 hours
Length of hospital stay | 30 days
  Days of hospital stay
Length of ICU stay | 30 days
  Days of ICU stay
Instrumental response | 30 days
  Changes in pulmonary echography
Proportion of adverse events | 30 days
  Rate of adverse events codified by Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Menichetti, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Richardson P, Griffin I, Tucker C, Smith D, Oechsle O, Phelan A, Rawling M, Savory E, Stebbing J. Baricitinib as potential treatment for 2019-nCoV acute respiratory disease. Lancet. 2020 Feb 15;395(10223):e30-e31. doi: 10.1016/S0140-6736(20)30304-4. Epub 2020 Feb 4. No abstract available. PMID 32032529
- [Result] Favalli EG, Biggioggero M, Maioli G, Caporali R. Baricitinib for COVID-19: a suitable treatment? Lancet Infect Dis. 2020 Sep;20(9):1012-1013. doi: 10.1016/S1473-3099(20)30262-0. Epub 2020 Apr 3. No abstract available. PMID 32251638